CLINICAL TRIAL: NCT01139359
Title: A Phase I Dose Escalation Study of Darinaparsin in Combination With CHOP in Previously Untreated Patients With Lymphomas Who Are Scheduled to Receive CHOP Alone
Brief Title: Safety Study of Darinaparsin in Combination With Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (CHOP) to Treat Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study enrollment was withdrawn as it is no longer the sponsor's intention to study this indication under this protocol.
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGL1003
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Lymphoma
Keywords: Lymphoma; Darinaparsin; CHOP; Frontline; PTCL; B-cell
MeSH Terms: conditions — Lymphoma | interventions — darinaparsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm, darinaparsin and CHOP (Experimental): open label, single arm, unblinded
  Interventions: Drug: darinaparsin; Drug: CHOP

INTERVENTIONS:
Drug: darinaparsin — I.V. darinaparsin given in a dose escalation manner, once a day for 5 days per cycle.
  Other Names: ZIO-101; Zinapar(TM)
Drug: CHOP — Cyclophosphamide 750 mg/m2 IV Day 8 of each Cycle; Doxorubicin 50 mg/m2 IV Day 8 of each Cycle; Vincristine 1.4 mg/m2 IV Day 8 of each Cycle; Prednisone 100 mg oral Days 8-12 of each Cycle.

SUMMARY:
This study is a Phase I trial of Darinaparsin in combination with CHOP for the treatment of lymphoma. Eligible patients will not have had any previous anti-cancer treatment and will be eligible to receive CHOP alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological or cytological confirmation of lymphoma who are previously untreated and are scheduled to receive CHOP alone. Since the objective of the study is the assessment of safety, eligible subjects may have any type of lymphoma (Hodgkin's or non-Hodgkin's, T-cell or B-cell), as long as the scheduled therapy is CHOP alone.
* Men and women of ≥18 years of age.
* ECOG performance score ≤2
* Life expectancy ≥12 weeks.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements, to be conducted <2 weeks prior to first dose of study drug:

  * Creatinine ≤1.5 × upper limit of normal (ULN) OR a calculated creatinine clearance ≥60 cc/min
  * Total bilirubin ≤2 × ULN
  * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤3 × ULN
  * Granulocytes in peripheral blood ≥1 × 109/L, hemoglobin ≥10 g/dL, and platelets ≥50,000 /µL
* Adequate vascular access for repeated blood sampling.
* Men and women of childbearing potential must agree to use effective contraception from Screening through 30 days after the last dose of study drug.
* Written informed consent in compliance with ZIOPHARM policies and the Human Investigation Review Committee (IEC/IRB) having jurisdiction over the site.

Exclusion Criteria:

* Arsenic allergy.
* New York Heart Association (NYHA) functional class ≥3 myocardial infarction (see Appendix 3) within 6 months.
* Myocardial dysfunction defined as scintigraphically- (MUGA [multiple gated acquisition scan], myocardial scintigram) or ultrasound-determined left ventricular ejection fraction (LVEF) <50%.
* Uncontrolled cardiac arrhythmia other than asymptomatic atrial fibrillation; a QTc ≥450 msec; or a ≥Grade 2 atrioventricular (AV) block or left bundle branch block (LBBB); or documented history of prolonged QTc.
* Pregnant and/or lactating women.
* Uncontrolled systemic infection (documented with microbiological studies).
* Metastatic brain or meningeal tumors. -Patients with seizure disorder requiring medication (such as anti- branch block (LBBB); or documented history of prolonged QTc.
* History of confusion or dementia or neurological condition that could mask a potential adverse response to the Study Drug, which may include transient ischemic attack, Parkinson's disease, thrombotic or hemorrhagic stroke, Alzheimer's, and other neurological disorders.
* Anticancer chemotherapy or immunotherapy for this indication.
* Radiotherapy during study or within 3 weeks of Study entry.
* Major surgery within 4 weeks of start of Study Drug dosing.
* Investigational drug therapy outside of this trial.
* History of invasive second primary malignancy diagnosed within the previous 3 years except for Stage I endometrial/cervical carcinoma or prostate carcinoma treated surgically, and non-melanoma skin cancer.
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of Study results.
* Any condition that is unstable or could jeopardize the safety of the patient and his/her compliance in the Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Define Toxicity profile | One Year
  This is an open-label, dose-escalation Phase I study to define the toxicity profile and the maximum tolerated dose (MTD) of intravenously administered darinaparsin in combination with CHOP in patients with previously untreated lymphomas who are scheduled to receive CHOP alone (rituximab is not permitted)
Maximum Tolerated Dose | One Year
  This is an open-label, dose-escalation Phase I study to define the toxicity profile and the maximum tolerated dose (MTD) of intravenously administered darinaparsin in combination with CHOP in patients with previously untreated lymphomas who are scheduled to receive CHOP alone (rituximab is not permitted).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan J. Lewis, MD, PhD, Study Director — ZIOPHARM, Oncology, Inc.